CLINICAL TRIAL: NCT06330623
Title: Developing Personalised, Relative Intensity Physical Activity Thresholds for Accelerometer-Derived Measures of Physical Activity in COPD (IMPACT)
Brief Title: Developing Personalised Relative Physical Activity Thresholds in COPD.
Acronym: IMPACT
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0929; 321895 (Other: HRA)
Record Dates: First submitted 2024-03-04; First posted 2024-03-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Absolute Intensity; Activity Monitors; Chronic Obstructive Pulmonary Disease; Exercise Capacity; Physical Activity; Relative Intensity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1 Cohort: These participants will be recruited from:
  * Previous research studies
  * COPD nursing ward
  * Pulmonary rehabilitation
- Phase 2 Cohort: These participants will be recruited from the pulmonary rehabilitation service.

SUMMARY:
The aim of this observational study is to translate the principle of individualised exercise prescription into the evaluation of daily absolute and relative intensity physical activity.

The main questions this study aims to answer are:

* Phase 1: What does physical activity (intensity) mean to people with COPD?
* Phase 2: Are there differences between time spent in absolute and relative physical activity for people with COPD?

Phase 1 Participants will take part in semi-structured interview (30-45 minutes) about living with COPD and perceptions of physical activity and how they perceive intensity. This will also include photovoice and photo-elicitation. Demographic information will be recorded and participants will also complete several respiratory symptom questionnaires.

Phase 2:

Participants will take part in physical activity testing before and after pulmonary rehabilitation while wearing physical activity monitors. Demographic information will be recorded and participants will also complete several respiratory symptom and physical activity questionnaires. Participants will also wear the physical activity monitors for 8 days after the pre-testing sessions and after their final pulmonary rehabilitation class.

Sub-study:

Participants will be asked to take images of barriers during physical activity, facilitators during physical activity, feelings during physical activity and types of physical activity they take part in for 8 days after their final pulmonary rehabilitation class. Participants will then take part in a semi-structured interview about the images their have taken while doing physical activity.

DETAILED DESCRIPTION:
Physical activity (PA) helps prevent and manage non-communicable diseases such as chronic obstructive pulmonary disease (COPD). Pulmonary rehabilitation (PR) has been shown to benefit people living with COPD by reducing breathlessness, increasing muscle strength, and improving the management of exacerbations. However, the improvement in PA in individuals with COPD remains inconsistent following PR. Despite the personalised nature of PA prescription during PR, the evaluation of free-living PA data has been limited to a 'one size fits all' approach using absolute intensity categories. Reduced exercise tolerance can result in PA being perceived at a high intensity relative to a person's exercise capacity, despite the absolute intensity being low. Exploring both the relative and absolute intensity of PA could offer additional insights and clinical relevance for the evaluation of physical activity in COPD populations.

The aim of this research is to translate the principle of individualised exercise prescription into the evaluation of daily absolute and relative intensity PA in a user-friendly format for PR teams and service users.

Phase 1 objective: To explore what PA means to people with COPD in the context of relative intensity and pulmonary rehabilitation.

Phase 2 objective: To examine the differences between time spent in physical activity intensity expressed in absolute and relative terms for people with COPD.

Phase 1: Semi-structured interviews will take place where participants will discuss their COPD and their perceptions of physical activity and relative intensity. The interviews will be in person (Biomedical research centre, Leicester) or over the phone/video call. The participants will complete several questionnaires about respiratory symptoms. Before taking part in the interviews, participants will also be asked to take pictures, using a camera provided, of when they are doing physical activity. This will be for a 7 day period before the interview.

Phase 2: Participants will take part in exercise testing and complete questionnaires pre and post pulmonary rehabilitation while wearing activity and gait monitors. Participants will also be asked to wear the activity monitors for 8-days after the pre-testing sessions and 8-days after their last pulmonary rehabilitation class. Following their last pulmonary rehabilitation class, 20 participants will be asked to take photographs during the period they are wearing accelerometers and motion sensors. When the participants return the devices, they will take part in an interview to discuss the images they have taken while taking part in physical activity.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Willing and able to provide informed consent for participation in the research.
* The patient has a confirmed diagnosis of COPD using spirometry (based on GOLD criteria (Agustí et al., 2023).
* Male or female, aged 40+ years
* Able to communicate in written and spoken English.

Exclusion Criteria:

* Unable to provide valid informed consent.
* Severe psychiatric disorders
* Aged less than 40 years
* Unable to understand written or spoken English.

Phase 2:

Inclusion Criteria:

* Willing and able to provide informed consent for participation in the research.
* The patient has a confirmed diagnosis of COPD using spirometry (based on GOLD criteria.
* The patient is referred for PR at the UHL.
* Male or female, aged 40+ years
* Able to communicate in written and spoken English

Exclusion Criteria:

* Unable to provide valid informed consent.
* Lack of motivation to participate in PR programme.
* Any-contra-indications absolute or relative to exercise training.
* Has had a cardiac event within last 6 weeks
* Severe psychiatric disorders
* Patients with a history of MRSA +ve screens (patients can be assessed and given an exercise programme but cannot attend the classes. Patients need to have 3 consecutive -ve MRSA swabs before they can attend).
* Aged less than 40 years
* Unable to understand written or spoken English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1:
  Patients from the COPD nursing ward, previous research studies and pulmonary rehabilitation programme.
  Phase 2:
  Patients from the pulmonary rehabilitation programme.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - Semi-structured Interviews | 30-45 minutes
  Semi-structured interview with individuals with COPD
Phase 2 - Differences between time spent in PA intensity expressed in absolute and relative intensity. | 8 days
  Differences between time spent in PA intensity expressed in absolute and relative using activity monitors (wrist and waist) for eight days before and after the PR programme.

SECONDARY OUTCOMES:
Phase 1 - Medical Research Council (MRC) Dyspnoea Scale | 2 minutes
  Medical Research Council (MRC) Dyspnoea Scale Minimum value: 1 Maximum value: 5 The higher the score, the worse the outcome (breathlessness).
Phase 1 - COPD Assessment Test (CAT) | 5 minutes
  COPD Assessment Test (CAT)
Phase 1 - Chronic Respiratory Questionnaire (CRQ-SR) | 5 minutes
  Chronic Respiratory Questionnaire (CRQ-SR)
Phase 1 - Photovoice and photo-elicitation | 7 days
  Photovoice is a qualitative research method that focuses on participants identifying and addressing important topics that matter to them through photography. This will gain greater insight from the participants about their experiences of participating in PA. Participant-generated images will be used to inform the photo-elicitation aspect of the interview to enable participants to capture in real time, more graphically illustrate their experiences and perceptions of different types of PA.
Phase 2 - Medical Research Council (MRC) Dyspnoea Scale | 2 minutes
  Medical Research Council (MRC) Dyspnoea Scale
Phase 2 - COPD Assessment Test (CAT) | 5 minutes
  COPD Assessment Test (CAT)
Phase 2 - Chronic Respiratory Questionnaire (CRQ-SR) | 5 minutes
  Chronic Respiratory Questionnaire (CRQ-SR)
Phase 2 - Gait Analysis | 45 minutes
  Gait Analysis - Speed, Variability, Asymmetry
Phase 2 - Exercise Capacity (ISWT) | 30-45 minutes
  Incremental Shuttle Walk Test
Phase 2 - Exercise Capacity (ESWT) | 15-30 minutes
  Endurance Shuttle Walk Test
Phase 2 - Clinical PROactive Physical Activity instrument in COPD (C-PPAC) | 5 minutes
  Clinical PROactive Physical Activity instrument in COPD (C-PPAC)
Phase 2 - Photovoice and photo-elicitation | 8 days
  Photovoice is a qualitative research method that focuses on participants identifying and addressing important topics that matter to them through photography. This will gain greater insight from the participants about their experiences of participating in PA. Participant-generated images will be used to inform the photo-elicitation aspect of the interview to enable participants to capture in real time, more graphically illustrate their experiences and perceptions of different types of PA.

CONTACTS AND LOCATIONS:
Overall Officials: University of Leicester University of Leicester, Principal Investigator — University of Leicester
Locations (1):
- NIHR Leicester Biomedical Research Centre - Respiratory, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data will only be available in publications.